CLINICAL TRIAL: NCT01907308
Title: A Phase II Single-arm Study of AMG 386 in Combination With Docetaxel for Advanced Urothelial Carcinoma After Failure of a Platinum-containing Regimen
Brief Title: Trebananib (AMG 386) in Combination With Docetaxel for Advanced Urothelial Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision to terminate the study
Sponsor: University of Colorado, Denver (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-1502.cc; NCI-2013-01348 (Other: National Cancer Institute)
Record Dates: First submitted 2013-07-16; First posted 2013-07-24 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Urothelial Carcinoma
Keywords: Bladder cancer; Urothelial cancer; Urothelial carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — trebananib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination of AMG 386 with Docetaxel (Experimental): All treated patients will receive AMG 386 30mg/kg IV weekly plus docetaxel 75mg/m2 IV every 3 weeks.
  Interventions: Drug: AMG 386; Drug: Docetaxel

INTERVENTIONS:
Drug: AMG 386 — Patients will receive AMG 386 30mg/kg IV weekly plus docetaxel 75mg/m2 IV every 3 weeks.
  Other Names: Trebananib
Drug: Docetaxel — Patients will receive AMG 386 30mg/kg IV weekly plus docetaxel 75mg/m2 IV every 3 weeks.
  Other Names: Docefrez; Taxotere

SUMMARY:
This study plans to learn more about the combination of AMG 386 and docetaxel for the treatment of advanced urothelial cancer. Subjects are being asked to be in this research study because they have advanced urothelial cancer which has progressed after treatment with a platinum-based therapy.

The hypothesis is that AMG 386 will increase the historical response rate of docetaxel as a single agent.

DETAILED DESCRIPTION:
AMG 386 is a medication made to stop the growth of blood vessels in cancer tissues. Cancer relies on new blood vessels to bring it oxygen and nutrients to grow. Docetaxel is currently approved by the FDA for advanced urothelial, hormone-refractory prostate, breast, non-small cell lung, gastric, and squamous cell carcinoma of the head and neck.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a histologically confirmed urothelial carcinoma. At least 50% of the tumor must demonstrate transitional cell histology.
2. Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
3. CT or MRI of the chest, abdomen, and pelvis, with or without contrast, within 28 days of registration. A whole body bone scan may be performed at the discretion of the treating physician.
4. Only if clinically indicated, a CT or MRI (MRI preferred) scan of the brain within 28 days of registration.
5. Progressive disease after a platinum-containing regimen (cisplatin or carboplatin) or intolerance to platinum-based therapy for urothelial carcinoma. Subjects who received adjuvant cisplatin or carboplatin-based chemotherapy for urothelial carcinoma and currently have recurrent or progressive disease are eligible.
6. Men or women > 18 years old
7. Generally well-controlled blood pressure with systolic blood pressure ≤ 140 mmHg AND diastolic blood pressure ≤ 90 mmHg prior to enrolment or randomization. The use of anti-hypertensive medications to control hypertension is permitted
8. Adequate organ and hematological function as evidenced by the following laboratory studies:

   a. Hematological function, as follows: i. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L ii. Platelet count ≥ 100 x 109/L iii. Hemoglobin ≥= 9 g/dL b. Hepatic function, as follows: i. Aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal (ULN), ii. Alanine aminotransferase (ALT) ≤ 2.5 x ULN iii. Alkaline phosphatase ≤ 2.0 x ULN iv. Total bilirubin within normal limits (WNL) c. Hemostatic function, as follows: i. International normalized ratio (INR) ≤ 1.5 ii. Activated Partial thromboplastin time (aPTT) ≤ 1.5 x ULN d. Renal function, as follows: i. Calculated creatinine clearance ≥ 40 cc/min according to the Cockcroft-Gault formula: Creatinine Clearance calculator (CrCl) (mL/min) = (140-age) x actual body weight (kg) (x 0.85 for females) 72 x serum creatinine (mg/dL) ii. Urinary protein quantitative value of ≤ 30 mg in urinalysis or ≤ 1+ on dipstick, unless quantitative protein is ≤ 1000 mg in a 24 hour urine sample e. Cardiac function, as follows (only in those with a known history of cardiac dysfunction or in those with symptoms indicative or cardiac dysfunction): i. Normal sinus rhythm or clinically stable arrhythmia well controlled on outpatient medication.

   ii. Left ventricular ejection fraction ≥ lower limit of normal (LLN) per institutional laboratory range, as determined by echocardiogram or multi gated acquisition scan (MUGA) scan within 28 days prior to enrollment. If no clear institutional standard, then the ejection fraction must be ≥ 50%.
9. All baseline laboratory results must be from within 14 days of registration
10. Competent to comprehend, sign, and date an institutional review board (IRB) - approved informed consent form
11. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
12. Subject plans to begin protocol-directed therapy within 7 days of registration
13. All patients will be offered enrollment in the correlative biomarkers study

Exclusion Criteria:

1. Three or more previous systemic therapies or combination regimens for urothelial carcinoma (e.g. cisplatin given with gemcitabine is considered one regimen) in the recurrent or metastatic setting.
2. Grade 2 or greater neuropathy
3. Known history of central nervous system metastases. An MRI or CT scan of the brain will be performed within 28 days of study enrollment.
4. History of arterial or venous thrombosis, including transient ischemic attack (TIA), within 12 months prior to enrollment
5. History of clinically significant bleeding within 6 months of study enrollment
6. Anticoagulation is allowed as long as the initiating thrombotic event was at least 12 months before enrollment. The use of aspirin and anti-platelet agents are also acceptable for any duration prior to enrollment. The concurrent use of low molecular weight heparin, heparinoids, or low dose warfarin (ie, 1 mg daily) for prophylaxis against thrombosis is acceptable while on study.
7. Subjects with pleural effusions or ascites.
8. Focal radiation therapy for palliation of pain from bony metastases within 21 days of study enrollment. Subjects who received radiation therapy must have recovered from all radiation induced toxicities prior to study enrollment
9. Currently or previously treated with AMG 386, or other molecules that inhibit the angiopoietins or Tie2 receptor including but not limited to, AZD-5180, XL-820, CEP 11981/SSR-106462, BSF-466,895, CGI-1842, LOC-590, XL-184, or CP- 8681596. (Previous treatment with bevacizumab is permitted.)
10. Current or previous treatment with docetaxel. (Previous treatment with paclitaxel is permitted.)
11. Treatment within 30 days prior to enrollment with strong immune modulators including but not limited to systemic cyclosporine, tacrolimus, sirolimus, mycophenolate mofetil, methotrexate, azathioprine, rapamycin, thalidomide, lenalidomide.
12. Clinically significant cardiovascular disease within 12 months prior to enrollment, including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, cerebrovascular accident, transient ischemic attack, congestive heart failure, or arrhythmias not controlled by outpatient medication
13. Major surgery within 28 days before study enrollment or still recovering from prior surgery
14. Minor surgical procedures, except placement of tunneled central venous access device within 3 days prior to enrollment/randomization.
15. Non-healing wound, ulcer (including gastrointestinal) or fracture
16. Pregnant (i.e., positive beta-human chorionic gonadotropin test) or current breast feeding
17. Subjects with a history of prior malignancy, except:

    * Malignancy treated with curative intent and with no known active disease present for > 3 years before enrollment and felt to be at low risk for recurrence by the treating physician.
    * Adequately treated non-melanomatous skin cancer or lentigo maligna without evidence of disease
    * Adequately treated cervical carcinoma in situ without evidence of disease
    * Prostatic intra-epithelial neoplasia without evidence of prostate cancer
18. Subject known to have tested positive for HIV or chronic hepatitis
19. Any condition which in the investigator's opinion makes the subject unsuitable for study participation
20. Female subject not consenting to the use of contraceptive method during the course of the study and for 6 months after administration of the last study medication
21. Subject currently is enrolled in or has not yet completed at least 30 days since ending other investigational device or drug study(s), or subject is receiving other investigational agent(s). Alternatively, for any recently administered investigational drugs, subjects may start treatment on this protocol after 4 half-lives of the previous investigational agent.
22. Subject has known sensitivity to any of the products to be administered during dosing (including any reaction to drugs formulated with polysorbate 80)
23. History of allergic reactions to bacterially produced proteins
24. Life expectancy of less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 21 days
  Determine the objective response rate (by RECIST 1.1 criteria) for the combination of AMG 386 (Trebananib) with docetaxel for the treatment of advanced or metastatic urothelial carcinoma, after failure of a platinum-containing regimen

SECONDARY OUTCOMES:
Overall survival | Up to 24 months
  Determine the overall survival for the combination of AMG 386 with docetaxel in advanced or metastatic urothelial carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Flaig, MD, Principal Investigator — Univerity of Colorado, Denver